CLINICAL TRIAL: NCT00370279
Title: Surgical Management of Pseudophakic and Aphakic Retinal Detachment; a Randomized Clinical Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8405
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2008-06-26 (Estimated); Status verified 2008-06

CONDITIONS: Pseudophakic Retinal Detachment; Aphakic Retinal Detachment
Keywords: Pseudophakic retinal detachment,; Aphakic retinal detachment,; Scleral buckling,; Primary vitrectomy,; Proliferative vitreoretinopathy
MeSH Terms: conditions — Vitreoretinopathy, Proliferative | interventions — Scleral Buckling

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- 1 (Active Comparator): scleral buckling
  Interventions: Procedure: scleral buckling, primary vitrectomy
- 2 (Active Comparator): Primary vitrectomy without encircling band
  Interventions: Procedure: scleral buckling, primary vitrectomy
- 3 (Active Comparator): Primary vitrectomy with encircling band
  Interventions: Procedure: scleral buckling, primary vitrectomy
- 4 (Active Comparator): Triamcinolone assisted vitrectomy
  Interventions: Procedure: scleral buckling, primary vitrectomy

INTERVENTIONS:
Procedure: scleral buckling, primary vitrectomy — Four different surgical techniques were performed(one in each arm); 1- scleral buckling, 2- primary vitrectomy without encircling band, 3- primary vitrectomy with encircling band, 4- triamcinolone assisted vitrectomy

SUMMARY:
To compare the visual and anatomical outcomes and complications of four surgical techniques (1- scleral buckling, 2- primary vitrectomy without encircling band, 3- primary vitrectomy with encircling band, 4- triamcinolone assisted vitrectomy) for management of pseudophakic and aphakic retinal detachment

ELIGIBILITY:
Inclusion Criteria:

* Cases of pseudophakic and aphakic retinal detachment with PVR grade A or B

Exclusion Criteria:

* PVR grade C
* History of surgery for RD
* Signs of diabetic retinopathy, AMD, glaucoma and macular hole
* History of ocular trauma
* Giant retinal tear

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-09

PRIMARY OUTCOMES:
Retinal reattachment rate
Visual acuity

SECONDARY OUTCOMES:
Proliferative vitreoretinopathy
Macular Pucker
Anisometropia
Choroidal detachment
Reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Ahmadieh, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Hamid Ahmadieh, MD, Tehran, Tehran Province, Iran